CLINICAL TRIAL: NCT05763238
Title: Effects of Pre-operative Exercise Therapy on Postoperative Outcomes in Children With Corrective Cardiac Surgeries.
Brief Title: Exercise Training in Children With Corrective Cardiac Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec/01386 Kanwal Zaheer
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Quality of Life; Congenital Heart Disease; Heart; Surgery, Heart, Functional Disturbance as Result
Keywords: Cardiopulmonary outcomes; Corrective cardiac surgeries; Preoperative Exercise therapy
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Preoperative Exercise therapy Patient Education, and post-operative conventional protocol.
  Interventions: Other: INTERVENTION GROUP
- Control group (Active Comparator): Patient Education, and post-operative conventional protocol.
  Interventions: Other: CONTROL GROUP

INTERVENTIONS:
Other: INTERVENTION GROUP — Preoperative Protocol:
  DAY 1: Incentive spirometry 1 set of 2 repetitions(each repetition includes 05 deep inhalations) 3 times a day.
  Active ROMS (3 sets of 5 repetitions of both upper and lower limb thrice a day) Walk, Static marching to 10 steps thrice a day. DAY 2: Incentive spirometry 1 set of 3 repetitions (each repetition includes 08-10 deep inhalation) 3 times a day.
  Active ROMS, 3 sets of 5 repetitions of both upper and lower limb thrice a day) Walk, Static marching to 15 steps thrice a day. DAY 3: Incentive spirometry,1 set of 3 repetitions(each repetition includes 10 deep inhalation) 3 times a day Active ROMS 3 sets of 5 repetitions of both upper and lower limbs thrice a day. Walk, Static marching to 20 steps thrice a day. Postoperative Protocol: Conventional protocol of respective cardiac setup
  Arms: Interventional Group
Other: CONTROL GROUP — Preoperative: Patients' parents will be educated about the disease process, surgery, it's possible complications, and precautions.
  Postoperative: Conventional protocol of respective cardiac setup
  Arms: Control group

SUMMARY:
To determine the effects of preoperative exercise therapy on postoperative cardiopulmonary outcomes and quality of life in children with corrective cardiac surgeries.Within literature there is limited evidence on preoperative exercise therapy in the pediatric population, positive results of the study can introduce a new tradition of preoperative exercise therapy and significantly reduce post-operative complications. Secondary complications would also be addressed in the study, a positive result can reduce the total costs by reducing hospital stays and improving the quality of life of child.

DETAILED DESCRIPTION:
Cardiac surgeries are often associated with some post-operative cardiopulmonary complications most often cardiac arrhythmias, pulmonary atelectasis, and hospital induced pneumonia and reduced inspiratory capacities which can be reduced by exercise therapy this study is therefore significant not only for the determination of the effects of preoperative exercise therapy, it will also provide a path toward pre-habilitation followed by effective postoperative cardiac rehabilitation which is mostly lacking in many setups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with congenital heart disease
* Undergoing elective corrective cardiac surgery
* Vitally stable

Exclusion Criteria:

* Having acquired heart disease or undergoing emergency cardiac surgeries
* Patients undergoing valvular repairing surgeries
* Functional status is limited due to conditions other than CHD or having any contraindications
* Inability to adhere to study protocols
* Participants who refused or withdrew from the study

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Health related Quality of life | 4 weeks
  Changes from pre-operative to 15 days after discharge from the hospital, measured through a Pediatric quality of life questionnaire consisting of 23 questions that are categorized into 4 major components namely, Physical functioning (8 items), Emotional functioning (5 items), Social functioning (5 items), School functioning (5 items). The scoring of the scale is based on the frequency of performance of particular activity ranging from 0 (mean never performed) to 5(mean always functioning).
Post-operative Pulmonary complications | 4 weeks
  Changes from pre-operative to post-operative, discharge day and 15 days after discharge from the hospital, measured through chest x-ray including Consolidation, Atelectasis, Pneumonitis, Pleural Effusion.
Abnormal heart rhythms | 7 days
  pre-operative to post-operative and discharge day observed through Electrocardiography (ECG) on cardiac monitor.
Forced Expiratory Volume in 1 second (FEV1) | 4 weeks
  Changes from pre-operative to post-operative, discharge day, and 15 days after discharge measured through the digital spirometer in Liters
Forced vital capacity | 4 Weeks
  Changes from pre-operative to post-operative, discharge day, and 15 days after discharge measured through the digital spirometer in Liters.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT(CPPT), Principal Investigator — Riphah International University
Locations (1):
- Armed forces institute of cardiology, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valkenet K, van de Port IG, Dronkers JJ, de Vries WR, Lindeman E, Backx FJ. The effects of preoperative exercise therapy on postoperative outcome: a systematic review. Clin Rehabil. 2011 Feb;25(2):99-111. doi: 10.1177/0269215510380830. Epub 2010 Nov 8. PMID 21059667
- [Background] Hulzebos EH, Smit Y, Helders PP, van Meeteren NL. Preoperative physical therapy for elective cardiac surgery patients. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD010118. doi: 10.1002/14651858.CD010118.pub2. PMID 23152283
- [Background] Bernier PL, Stefanescu A, Samoukovic G, Tchervenkov CI. The challenge of congenital heart disease worldwide: epidemiologic and demographic facts. Semin Thorac Cardiovasc Surg Pediatr Card Surg Annu. 2010;13(1):26-34. doi: 10.1053/j.pcsu.2010.02.005. PMID 20307858